CLINICAL TRIAL: NCT05403931
Title: The Effectiveness of Low Level Laser Therapy on Particular Joint Points and Acupuncture Points on Knee Joints in Grade III Knee Osteoarthritis
Acronym: LLLT OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Teknologi Malaysia (Other)
Responsible Party: Principal Investigator, Adnan Afzal, Principal Investigator, Universiti Teknologi Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Admin/GDEC/276/20
Record Dates: First submitted 2022-05-06; First posted 2022-06-03 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Interventional study to compare the effectiveness of low level laser therapy on two groups of points of irradiation in knee OA grade III. One group of points involves 6-7 particular points on tibiofemoral and patellofemoral joints. Other group involves the 6-7 particular acupuncture points which have been previously used in a study. Outcomes will indicate that which group irradiation will produce better therapeutic results.
Who Masked: Outcomes Assessor
Masking Description: Person assessing the outcomes will have no knowledge that patient received laser therapy on which points of knee area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Particular joint point group (Experimental): This group will receive laser irradiation on 6-7 particular points including 4-5 on tibiofemoral and 2 on patellofemoral joint.
  Interventions: Device: Low level laser therapy
- Acupuncture points group (Experimental): This group will receive laser irradiation on 6-7 particular acupuncture points which have been previously used in another study and or identified in literature.
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: Low level laser therapy — Omega XP is the particular device producing low level laser therapy and has been in use for therapeutic purposes to treat different musculoskeletal conditions.
  Other Names: Cold laser therapy

SUMMARY:
LLLT is in use to treat different musculoskeletal condition. Osteoarthritis is one of the conditions needing LLLT for therapeutic effects. LLLT has been used in different previous studies using different points on joint and also on acupuncture points. This study is going to compare the effectiveness of LLLT on both points. Omega xp device is going to be used in this study.

DETAILED DESCRIPTION:
LLLT is a non-invasive modality to treat variety of musculoskeletal conditions. Photobiomodulation has been studies for last two decades in different perspectives and on different musculoskeletal condition. Studies suggest profound results due to effect of LLLT at the cellular level. Osteoarthritis is one of the most common debilitating musculoskeletal condition affecting people worldwide. Statistics indicate an increase in this debilitating condition in future. Knee OA is more common amongst other OA of the body. LLLT has been used in previous studies to see the impact on pain and functional performance in knee OA. LLLT has been used on different points on knee joint and also applied on acupuncture points of the knee joints. Different outcomes were used to assess LLLT effectiveness including pain, ROM and even different biomarkers. This study is going to use LLLT on different particular joint points of knee and also acupuncture points of the knee joint and compare the outcomes. This study will present evidence for the clinicians to use LLLT on either the particular joint points or acupuncture points for better clinical outcomes.

ELIGIBILITY:
* Inclusion Criteria:

  * Pain in the knee joint ( minimum 30/100 on VAS )
  * Kellgren-Lawrence Grade III knee OA
  * ACR criteria for knee OA with radiological findings including ;

    * age 35 and above
    * joint crepitus
    * less than 30 minutes of morning stiffness
* Exclusion Criteria:

  * Knee OA grade other than III.
  * Any contraindication of LLLT including;

    * pregnancy
    * carcinoma involving knee area
  * Steroids and NSAIDS use

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index ( WOMAC ) | Baseline
  Western Ontario and McMaster University Osteoarthritis Index is a standard questionnaire used in knee OA to assess the outcome of an intervention. It's 24 items scale which covers pain, stiffness and function. The score ranges from 0-96. 0 means the best health or best performance and 96 is the worst health status or performance.
Western Ontario and McMaster University Osteoarthritis Index ( WOMAC ) | 2nd week
  Western Ontario and McMaster University Osteoarthritis Index is a standard questionnaire used in knee OA to assess the outcome of an intervention. It's 24 items scale which covers pain, stiffness and function. The score ranges from 0-96. 0 means the best health or best performance and 96 is the worst health status or performance.
Western Ontario and McMaster University Osteoarthritis Index ( WOMAC ) | 3rd week
  Western Ontario and McMaster University Osteoarthritis Index is a standard questionnaire used in knee OA to assess the outcome of an intervention. It's 24 items scale which covers pain, stiffness and function. The score ranges from 0-96. 0 means the best health or best performance and 96 is the worst health status or performance.
Western Ontario and McMaster University Osteoarthritis Index ( WOMAC ) | 4th week
  Western Ontario and McMaster University Osteoarthritis Index is a standard questionnaire used in knee OA to assess the outcome of an intervention. It's 24 items scale which covers pain, stiffness and function. The score ranges from 0-96. 0 means the best health or best performance and 96 is the worst health status or performance.
Western Ontario and McMaster University Osteoarthritis Index ( WOMAC ) | 16th week
  Western Ontario and McMaster University Osteoarthritis Index is a standard questionnaire used in knee OA to assess the outcome of an intervention. It's 24 items scale which covers pain, stiffness and function. The score ranges from 0-96. 0 means the best health or best performance and 96 is the worst health status or performance.
Timed Up and Go test ( TUG ) | Baseline
  Timed Up and Go test assesses the balance and is widely used in the clinical outcomes assessment. It's measured in seconds. Lesser the time means good balance and longer the time means poor balance.
Timed Up and Go test ( TUG ) | 2nd week
  Timed Up and Go test assesses the balance and is widely used in the clinical outcomes assessment. It's measured in seconds. Lesser the time means good balance and longer the time means poor balance.
Timed Up and Go test ( TUG ) | 3rd week
  Timed Up and Go test assesses the balance and is widely used in the clinical outcomes assessment. It's measured in seconds. Lesser the time means good balance and longer the time means poor balance.
Timed Up and Go test ( TUG ) | 4th week
  Timed Up and Go test assesses the balance and is widely used in the clinical outcomes assessment. It's measured in seconds. Lesser the time means better performance and longer the time means poor performance.
Timed Up and Go test ( TUG ) | 16th week
  Timed Up and Go test assesses the balance and is widely used in the clinical outcomes assessment. It's measured in seconds. Lesser the time means good balance and longer the time means poor balance.
Visual Analog Scale ( VAS ) | Baseline
  Visual Analog Scale is a widely used tool to assess pain in knee OA. The score ranges from 0-100. 0 means no pain and 100 means the worst pain.
Visual Analog Scale ( VAS ) | 2nd week
  Visual Analog Scale is a widely used tool to assess pain in knee OA. The score ranges from 0-100. 0 means no pain and 100 means the worst pain.
Visual Analog Scale ( VAS ) | 3rd week
  Visual Analog Scale is a widely used tool to assess pain in knee OA. The score ranges from 0-100. 0 means no pain and 100 means the worst pain.
Visual Analog Scale ( VAS ) | 4th week
  Visual Analog Scale is a widely used tool to assess pain in knee OA. The score ranges from 0-100. 0 means no pain and 100 means the worst pain.
Visual Analog Scale ( VAS ) | 16th week
  Visual Analog Scale is a widely used tool to assess pain in knee OA. The score ranges from 0-100. 0 means no pain and 100 means the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Afzal, PhD, Principal Investigator — University of Technology Malaysia
Locations (1):
- Central Park Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hegedus B, Viharos L, Gervain M, Galfi M. The effect of low-level laser in knee osteoarthritis: a double-blind, randomized, placebo-controlled trial. Photomed Laser Surg. 2009 Aug;27(4):577-84. doi: 10.1089/pho.2008.2297. PMID 19530911
- [Background] Bjordal JM, Couppe C, Chow RT, Tuner J, Ljunggren EA. A systematic review of low level laser therapy with location-specific doses for pain from chronic joint disorders. Aust J Physiother. 2003;49(2):107-16. doi: 10.1016/s0004-9514(14)60127-6. PMID 12775206
- [Background] Al Rashoud AS, Abboud RJ, Wang W, Wigderowitz C. Efficacy of low-level laser therapy applied at acupuncture points in knee osteoarthritis: a randomised double-blind comparative trial. Physiotherapy. 2014 Sep;100(3):242-8. doi: 10.1016/j.physio.2013.09.007. Epub 2013 Nov 15. PMID 24418801